CLINICAL TRIAL: NCT02001831
Title: Effect of a Nutrition Supplement Containing Fish Oil, Whey Protein, Vitamin D, and Resveratrol, on Muscular and Cognitive Function in Older Adults
Brief Title: Multi-ingredient Nutrition Supplement in Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University College Dublin (Other)
Collaborators: Smartfish AS (Industry)
Responsible Party: Principal Investigator, Brendan Egan, Lecturer in Sport and Exercise Science, University College Dublin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SMF-3000
Record Dates: First submitted 2013-08-15; First posted 2013-12-05 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-11

CONDITIONS: Physical Disability
Keywords: Sarcopenia; Frailty; Aging; Skeletal muscle; Nutrition
MeSH Terms: conditions — Sarcopenia; Frailty | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supplement (Experimental): Liquid nutrient support (quantity 200 mL per day; energy 200 kcal per day):
  Carbohydrate 28.5 g
  Protein 8 g as Whey Protein Isolate
  ω-3 PUFA 3000 mg, as DHA 1500mg, as EPA 1500mg
  Vitamin D3 10 μg
  Resveratrol 150 mg
  Interventions: Dietary Supplement: Supplement
- Control (Placebo Comparator): Placebo control
  Liquid nutrient support
  Quantity 200 mL per day - fruit juice only i,e. in absence of bioactives present in the "supplement" (whey protein, omega 3, vitamin D and resveratrol).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Supplement
  Arms: Supplement
Dietary Supplement: Placebo
  Arms: Control

SUMMARY:
The aims of the present study are:

i. To conduct a population study of body composition, muscle function and ability to undertake activities of daily living in elderly Irish individuals

ii. To investigate the effect of a six month period of nutrition supplement support on lean tissue mass, and muscle and cognitive function in individuals aged 70 to 80 years.

DETAILED DESCRIPTION:
The study is a population study and 6 month randomised control trial (RCT) of men and women aged 70 to 80. The supplement and placebo will be provided in the form of a small 200 mL sealed TetraPak carton and is presented in a highly-palatable, juice-based (pomegranate and apple) formulation. The study groups (n=25 per group) for the RCT are:

Control - a control group receiving a placebo nutrient support (200 mL juice; energy ~ 100 kcal per day)

Supplement - a nutrient group receiving a liquid nutrient support (quantity 200 mL per day; energy 200 kcal per day):

Carbohydrate 28.5 g Protein 8 g as Whey Protein Isolate (i) ω-3 PUFA (ii) 3000 mg, as DHA 1500mg, as EPA 1500mg Vitamin D3 (iii) 10 μg Resveratrol (iv) 150 mg

(i) Whey protein isolate - increasing protein intake in elderly individuals is widely proposed as key preventing the decline in muscle mass with aging, (ii) ω-3/EPA/DHA fatty acids - increasing ω-3 consumption is associated with improvements in inflammatory status, blood lipid profile and cognitive function in various populations (iii) A relative deficiency in vitamin D is widely reported in Western populations, whereas recent reports have suggested vitamin D3 supplementation as efficacious for muscle function, (iv) Resveratrol, a polyphenol derived from grape skin that shows promise as a supplement to improve muscle function, metabolic health, prevent wasting and promote longevity.

Participants will undertake a first preliminary screening, which will take part at the Human Performance Laboratory at the University College Dublin (UCD) Institute for Sport and Health, or, alternatively, in a home-based environment, according to participants preferences, in order to assess inclusion/exclusion criteria.

After having examined the participant information leaflet, participants will provide informed consent in writing, complete the medical history examination, a food intake diary and food frequency questionnaire as well as habitual physical activity level questionnaire (CHAMPS).

Next, they will have their stature, body composition, and functional capacity assessed as described below. If fulfilling the eligibility criteria, subjects will undertake 3 assessment sessions (at baseline, 12 wk & 24 wk) at the Human Performance Laboratory at the UCD Institute for Sport and Health, consisting of body composition, functional capacity, and cognitive performance assessment.

In detail:

i. Body composition (fat, muscle and bone mass by Dual Energy X-Ray Absorptiometry (DXA) (Expected time ~ 15 min)

ii. Provide a blood sample taken via venepuncture to a superficial antecubital vein to be later analysed to assess lipidemic profile, plasma glucose, insulin, and inflammatory markers (Expected time ~ 5 min)

iii. Measurement of muscle strength and lower extremity muscle function in simulated activities of daily living by hand grip, usual walking speed, chair rise test, sit and reach test, and balance test [Short Performance Battery Test (Guralnik et al. 1994)]. (Expected time ~ 40 min)

iv. Assessment of cognitive function by the following battery modeled upon that used in Witte et al. (2013) (Expected time ~ 45 min):

* Timed Up and Go test
* Trail Making Test (TMT) part A and B
* Auditory Verbal Learning Test
* Stroop Colour-Word Test
* Verbal Fluency
* Forward and Backward Digit Spans
* Cognitive Failures Questionnaire

ELIGIBILITY:
Inclusion Criteria:

* ≥ 70 years of age
* Medically stable, according to Greig et al. (1994)
* BMI between 20 and 30 kg/m2
* Sedentary lifestyle, defined by ≤125 min/week of activity on the CHAMPS-18 questionnaire;

Exclusion criteria:

* Not medically stable by Greig criteria, and the medical history details in the ethics form
* Conducting an active lifestyle
* Skeletal muscle index (SMI) of ≥ 6.75 kg/m2 for women or ≥ 10.75 kg/m2 for men according to Janssen et al. (2003)
* Cognitive impairment expressed as mini mental state examination (MMSE) score ≤ 23.
* Current or recent (8 wk) use of fish-oil supplement intake
* Current or recent (8 wk) use of proteins, vitamins or other supplements interfering the metabolic scope

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-08 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Total and appendicular muscle mass | Change from Baseline at day 84 & day 168
  By means of measurement of lean body mass using dual-energy X-ray absorptiometry (DXA)

SECONDARY OUTCOMES:
Lower extremity physical function | Change from Baseline at day 84 & day 168
  By means of score ranging from 0 (worst performance) to 12 (best performance) achieved on the Short Performance Battery Test (Guralnik et al J Gerontol. 1994 49(2):M85-94)
Cognitive performance | Change from Baseline at day 84 & day 168
  By means of performances in the following battery: Timed Up and Go test, Trail Making Test (TMT) part A and B, Auditory Verbal Learning Test, Stroop Colour-Word Test, Verbal Fluency, Forward and Backward Digit Spans, and Cognitive Failures Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe De Vito, MD, PhD, Study Director — School of Public Health, Physiotherapy and Population Sciences. University College Dublin
Locations (1):
- UCD Institute for Sport and Health, Dublin, Ireland

REFERENCES:
- [Background] Greig CA, Young A, Skelton DA, Pippet E, Butler FM, Mahmud SM. Exercise studies with elderly volunteers. Age Ageing. 1994 May;23(3):185-9. doi: 10.1093/ageing/23.3.185. PMID 8085501
- [Background] Janssen I, Baumgartner RN, Ross R, Rosenberg IH, Roubenoff R. Skeletal muscle cutpoints associated with elevated physical disability risk in older men and women. Am J Epidemiol. 2004 Feb 15;159(4):413-21. doi: 10.1093/aje/kwh058. PMID 14769646
- [Background] Witte AV, Kerti L, Hermannstadter HM, Fiebach JB, Schreiber SJ, Schuchardt JP, Hahn A, Floel A. Long-chain omega-3 fatty acids improve brain function and structure in older adults. Cereb Cortex. 2014 Nov;24(11):3059-68. doi: 10.1093/cercor/bht163. Epub 2013 Jun 24. PMID 23796946
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Derived] Moran C, Scotto di Palumbo A, Bramham J, Moran A, Rooney B, De Vito G, Egan B. Effects of a Six-Month Multi-Ingredient Nutrition Supplement Intervention of Omega-3 Polyunsaturated Fatty Acids, vitamin D, Resveratrol, and Whey Protein on Cognitive Function in Older Adults: A Randomised, Double-Blind, Controlled Trial. J Prev Alzheimers Dis. 2018;5(3):175-183. doi: 10.14283/jpad.2018.11. PMID 29972210